CLINICAL TRIAL: NCT02022761
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose, Phase I Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Inhaled Laninamivir Octanoate in Adults With Chronic Asthma
Brief Title: Safety, Tolerability and Pharmacokinetics of Inhaled Laninamivir Octanoate TwinCaps® DPI in Adults With Chronic Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biota Scientific Management Pty Ltd (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: Vaxart (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BTA51-350-101
Record Dates: First submitted 2013-12-22; First posted 2013-12-30 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Asthma
Keywords: Mild or moderate asthmatics; Adults; Laninamivir
MeSH Terms: conditions — Asthma; Lymphoma, Follicular | interventions — laninamivir; CS 8958

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 40 mg Laninamivir octanoate (Experimental): Dry Powder Inhaler
  Interventions: Drug: Laninamivir octanoate
- 80 mg Laninamivir octanoate (Experimental): Dry Powder Inhaler
  Interventions: Drug: Laninamivir octanoate
- Matching placebo (Placebo Comparator): Dry Powder Inhaler
  Interventions: Drug: Laninamivir octanoate

INTERVENTIONS:
Drug: Laninamivir octanoate — 40 mg dose consists of 2 laninamivir octanoate TwinCaps® DPI 80 mg dose consists of 4 laninamivir octanoate TwinCaps® DPI (2 administered 12 hours apart)
  Other Names: CS-8958

SUMMARY:
This is a single centre, randomized, double-blind, placebo-controlled, single ascending dose study, in which the safety and pharmacokinetics of laninamivir octanoate administered by inhalation via the TwinCaps® DPI will be assessed in adults with mild or moderate chronic asthma.

DETAILED DESCRIPTION:
32 subjects, as two sequential groups of 16 subjects at each dose level (40 mg and 80 mg), will be randomised 3:1 to receive active drug or matching placebo.

Males and females aged 18 to 65 years inclusive, with mild or moderate chronic asthma.

Stratum 1: Mild asthma - requiring treatment consistent with Global Initiative for Asthma (GINA) Step 2 Stratum 2: Moderate asthma - requiring treatment consistent with GINA Step 3

Following a screening period of up to 30 days, eligible consenting subjects will be admitted to the clinic on the morning of Day 1. Laninamivir octanoate will be administered on Day 1. Subjects will remain in the clinic until Day 3 and will return for subsequent outpatient visits on Day 5, Day 6 and Day 7. A final follow-up visit for safety evaluations will occur on Day 14 ± 1 (or at the time of premature discontinuation). Each subject will participate in the study for approximately 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects 18 to 65 years of age, inclusive
2. Body mass index (BMI) within the range of 19.0 to 33.0 kg/m2, inclusive at screening
3. Minimum weight of 55.0 kg at screening and pre-dose Day 1
4. Clinical diagnosis of asthma by a physician for ≥12 months prior to screening confirmed in writing and/or by medical records
5. Mild asthmatics currently requiring treatment with low dose inhaled corticosteroids or other low intensity treatment OR Moderate asthmatics, requiring treatment with low dose inhaled corticosteroids and long-acting beta agonists, medium- high dose inhaled corticosteroids alone or low dose inhaled corticosteroids and other low intensity treatment8
6. Well controlled asthma for 1 month prior to dosing defined by the following:

   1. Daytime symptoms occur ≤8 times/ 4 weeks
   2. Daily activity is not limited by asthma
   3. No nocturnal symptoms resulting in nighttime awakenings
   4. Use of short-acting beta-agonist (SABA) ≤8 times/4 weeks for the treatment of symptoms
7. There has been no change in asthma medication (dose or regimen) within 4 weeks prior to dosing
8. Pre-short-acting β2 agonist (SABA) forced expiratory volume in 1 second (FEV1) of ≥80% of predicted normal values at screening
9. Non-smokers for at least 6 months prior to screening and agrees not to smoke during the study
10. Negative test results for smoking status at screening (urine cotinine) and pre-dose Day 1 (Smokerlyser)
11. Female subjects of childbearing potential must be practising true abstinence when this is in line with the preferred and usual lifestyle of the subject (Periodic abstinence, e.g. calendar, ovulation, symptothermal, post-ovulation methods and withdrawal are not acceptable methods of contraception), or be using and willing to continue using a medically acceptable form of birth control for at least 1 month prior to screening (at least 3 months for hormonal contraceptives) and for at least 1 month after the last study drug administration
12. Male subjects of reproductive potential who are not truly abstinent must be using and willing to continue using medically acceptable contraceptive precautions from screening and for at least 1 month after the last study drug administration
13. Female subjects must have a negative serum pregnancy test at screening and a negative urine pregnancy test pre-dose Day 1
14. Able to speak, read, and understand English sufficiently to understand the nature of the study, to provide informed consent, and to allow completion of all study assessments
15. Must provide written informed consent prior to the initiation of any protocol-specific procedures

Exclusion Criteria:

1. A history of a life-threatening asthma exacerbation that required intubation and mechanical ventilation
2. History of severe asthma exacerbation in the last year that required the use of systemic corticosteroids (tablets, suspension or injection)
3. Hospitalization or a visit to ER because of asthma in the last year
4. Intensive care admission for asthma in the previous 5 years
5. Any clinically significant abnormalities on clinical chemistry, haematology, or urinalysis, as judged by the investigator (at screening and/or Day -1)
6. Clinically significant abnormalities on physical examination, medical history, 12-lead ECG, or vital signs, as judged by the investigator (at screening or pre-dose Day 1)
7. A QTcF >430 msec for male subjects and >450 msec for female subjects on ECG at screening or pre-dose Day 1
8. History or presence of any clinically significant illness (e.g., cardiovascular, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, musculoskeletal, or psychiatric) or any other condition, which in the opinion of the investigator would jeopardize the safety of the subject or the validity of the study results
9. History or clinical evidence of other respiratory disease (e.g., COPD, cystic fibrosis)
10. Recent (within 2 weeks) or current signs or symptoms of a respiratory infection at screening or pre-dose Day 1
11. Currently taking theophylline or has taken theophylline in the 3 months prior to screening
12. Use of non-prescription drugs within 3 days prior to Day 1
13. Use of prescription medications (except acceptable asthma medications, acceptable forms of birth control, and hormone replacement) and recreational drugs within 14 days prior to Day 1
14. Positive urine drug screen or breath alcohol test at screening or pre-dose Day 1
15. Female subjects who are pregnant or lactating or who are planning to become pregnant within 30 days of study drug administration
16. History of allergy, hypersensitivity, or serious adverse reaction to lactose or neuraminidase inhibitors
17. Previous exposure to laninamivir octanoate
18. Positive for Hepatitis B surface antigen, Hepatitis C virus antibody, or Human Immunodeficiency Virus (HIV) p24 antigen/antibodies at screening
19. Donation or loss of ≥500 mL whole blood within 2 months prior to Day 1
20. Current or pending legal charges or currently on probation, based on subject report
21. Receipt of an investigational product in a clinical trial within 30 days or 5 half-lives, whichever is longer, prior to Day 1
22. Concurrent enrolment in any other type of medical research, judged by the investigator not to be scientifically or medically compatible with this study
23. An employee of the sponsor or research site personnel directly affiliated with this study or their immediate family members defined as a spouse, parent, sibling, or child, whether biological or legally adopted
24. A subject who, in the opinion of the investigator, is not considered to be suitable and is unlikely to comply with the study protocol for any reason

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-10; Primary Completion 2013-10 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of single ascending doses (40 mg and 80 mg) of laninamivir octanoate administered by inhalation via the TwinCaps® DPI in adults with mild or moderate chronic asthma. | Subjects assessed at clinic visits and up to 14 days post-dose
  Safety and tolerability data will be presented according to the dose group and asthma Strata. All safety data will be summarized with descriptive statistics and included assessments of SAEs, AEs, Laboratory Results, Vital Signs, ECGs, Spirometry parameters, Con Meds, Physical Exam findings

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics of laninamivir octanoate and its active metabolite laninamivir following administration of 40 mg & 80 mg doses of laninamivir octanoate by inhalation via the TwinCaps® DPI in adults with mild or moderate chronic a | Samples are collected up to 144 hours post-dose
  Cohort 1 - Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 96, 120 and 144 hours post dose Cohort 2 - Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 12.5, 13, 13.5, 14, 15, 16, 18, 20, 24, 36, 48, 96, 120 and 144 hours post dose
  Pharmacokinetic concentration data and PK parameters will be calculated and summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Jolanta Airey, Dr, Study Director — Biota Scientific Management Pty Ltd
Locations (1):
- Respiratory Clinical Trials, London, United Kingdom